CLINICAL TRIAL: NCT03479996
Title: Evaluation of Postoperative Pain After Tension-free Obturator Tape Operation (TVT-O) With or Without Local Anesthetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, ofer gemer, Director of gynecological surgery, BMC, Barzilai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRZ 0005-18 CTIL
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anesthetic (Experimental)
  Interventions: Drug: Marcaine 0.5 % Injectable Solution
- Control (No Intervention)

INTERVENTIONS:
Drug: Marcaine 0.5 % Injectable Solution — Intra -operative injection into obturator membrane
  Arms: Anesthetic

SUMMARY:
BACKGROUND:

Compare the pain intensity after TVT-O procedure in the inner part of the thigh where the anesthetic substance will be injected versus the inner part of of the thigh without anesthetic injection in the same woman.

The advantage of this work is that this method of testing neutralizes the effect of pain thresholds of different women.

If an advantage will be found in injecting anesthetic as a reduction in postoperative pain, it could be recommended for all women who undergo surgery of this kind.

METHODS:

Preoperative women will be offered the opportunity to participate in the study after a detailed explanation of the study and determine a date for an elective TVT-O procedure. After signing the Informed Consent Form, they will undergo a TVT-O procedure with injection of anesthetic into one of the obturators membranes. In a random order, Marcaine 5-ml will be injected into a left or right obturator membrane.

One side with Marcaine (Bupivacaine HCL) 0.5% 5 mg / mL Injection,opposite side without injection of any anesthetic.

Before and after surgery, patients will receive Visual Analogue Scale (VAS) instruction and will be polled at the following time points: 1,6,12,24 hours after surgery per inner part of the thigh separately. Each patient will rate the intensity of the pain she feels on the pain questionnaire at each of the time points mentioned before.

ELIGIBILITY:
Inclusion Criteria:

• Women undergoing TVT-O

Exclusion Criteria:

• Repeat surgery

Ages: 35 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Leg pain | 1 hour after surgery
  VAS score
Leg pain | 6 hours after surgery
  VAS score
Leg pain | 12 hours after surgery
  VAS score
Leg pain | 24 hours after surgery
  VAS score

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Gemer, Prof., Principal Investigator — Barzilai Medical Center
Locations (1):
- Barzilay University Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latthe PM, Foon R, Toozs-Hobson P. Transobturator and retropubic tape procedures in stress urinary incontinence: a systematic review and meta-analysis of effectiveness and complications. BJOG. 2007 May;114(5):522-31. doi: 10.1111/j.1471-0528.2007.01268.x. Epub 2007 Mar 16. PMID 17362484
- [Background] Cheng D, Liu C. Tension-free vaginal tape-obturator in the treatment of stress urinary incontinence: a prospective study with five-year follow-up. Eur J Obstet Gynecol Reprod Biol. 2012 Apr;161(2):228-31. doi: 10.1016/j.ejogrb.2012.01.011. Epub 2012 Feb 13. PMID 22336228
- [Background] Duckett J, Baranowski A. Pain after suburethral sling insertion for urinary stress incontinence. Int Urogynecol J. 2013 Feb;24(2):195-201. doi: 10.1007/s00192-012-1863-3. Epub 2012 Jul 3. PMID 22752013
- [Background] Hazewinkel MH, Hinoul P, Roovers JP. Persistent groin pain following a trans-obturator sling procedure for stress urinary incontinence: a diagnostic and therapeutic challenge. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Mar;20(3):363-5. doi: 10.1007/s00192-008-0714-8. Epub 2008 Sep 4. PMID 18769847
- [Background] Tommaselli GA, Di Carlo C, Formisano C, Fabozzi A, Nappi C. Effect of local infiltration analgesia on post-operative pain following TVT-O: a double-blind, placebo-controlled randomized study. Arch Gynecol Obstet. 2014 Aug;290(2):283-9. doi: 10.1007/s00404-014-3186-8. Epub 2014 Mar 6. PMID 24599566
- [Derived] Volchok V, Kapustian V, Namazov A, Zangen R, Anteby EY, Gemer O. Intra-obturator bupivacaine injection and post-operative pain following the trans-obturator tension-free vaginal tape procedure: randomized study. Arch Gynecol Obstet. 2024 Jun;309(6):2937-2941. doi: 10.1007/s00404-024-07533-y. Epub 2024 May 14. PMID 38743075